CLINICAL TRIAL: NCT04392947
Title: Treatment of Major Depressive Disorder With Bilateral Theta Burst Stimulation
Acronym: TBS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government); Institute of Clinical Epidemiology and applied Biometry, University Tuebingen, Germany (Unknown); Center of Clinical Trials, University Tuebingen, Germany (Unknown); University of Ulm (Other); Department of Psychiatry and Psychotherapy, University Regensburg, Germany (Unknown); Department of Psychiatry and Psychotherapy, University Wuerzburg, Germany (Unknown); Department of Psychiatry and Psychotherapy, University Munich (LMU), Germany (Unknown); Department of Psychiatry and Psychotherapy, University Leipzig, Germany (Unknown); Department of Psychiatry, Psychotherapy and Psychosomatics, Medical Faculty, University of Augsburg, Bezirkskrankenhaus Augsburg, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01KG2003 BMBF
Record Dates: First submitted 2020-05-08; First posted 2020-05-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder
Keywords: major depression; theta burst stimulation; dorsolateral prefrontal cortex; randomized; sham-controlled; multicenter
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The usage of a special active/placebo (A/P) coil in combination with an electrical co-stimulation will guarantee masking.
  A hard cover surrounds the A/P coil and for this reason it is not possible to see which side is the active side of the coil. By entering a randomized code into the stimulator, the operator receive information whether the coil is in the correct position or has to be flipped around. The code does not allow third parties to identify to which study arm a patient has been assigned. The concealment of the assignment remains until the statistical analysis is finished.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- combined iTBS/cTBS (Active Comparator): Combined theta burst stimulation (TBS) of the left (intermittent TBS, iTBS) and right (continuous TBS, cTBS) dorsolateral prefrontal cortex (dlPFC; F3 and F4 according to EEG10/20 system). Each stimulation session will comprise 2 trains of 600 stimuli each applied in bursts of three pulses at 50 Hz given every 200 ms. iTBS will be applied 20 times for 2 s every 10 s. In the same session, stimulation with cTBS will be applied continuously for 40 s. Intensity of iTBS/cTBS will be standardized at 80 % of the resting motor threshold (rMT).
  Additionally, patients receive an electrical co-stimulation of the forehead. One electrode is fixed to FZ and the 2nd one is either fixed to the left forehead (iTBS) or the right forehead (cTBS), rectangular aligned to the upper edge of the FZ-electrode with a distance of 0.5 cm. Intensity of the co-stimulation is applied with 50% of TBS-intensity.
  Interventions: Device: Transcranial Magnetic Stimulation
- sham stimulation (Sham Comparator): Setup is identical to combined active iTBS/cTBS but TBS is not actively delivered
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — MagVenture Coil Cool B70 A/P
  Arms: combined iTBS/cTBS
Device: Sham Transcranial Magnetic Stimulation — MagVenture Coil Cool B70 A/P without TMS being actively delivered
  Arms: sham stimulation

SUMMARY:
This is a randomized, double-blind, sham-controlled multicenter clinical trial. The aim is to provide evidence for efficacy of TBS in the treatment of patients with major depression. There will be a direct comparison between combined cTBS/iTBS with sham TBS. Overall, 236 patients with major depression will be randomized either to active TBS or sham TBS in a 1:1 ratio. The planned stimulation paradigms will be applied as add-on therapy to standard therapy (antidepressive medication and / or psychotherapy). Patients will receive 30 stimulation sessions in a 6-week treatment period (one session daily from Monday to Friday). Follow up assessments are scheduled 1 and 3 months after end of treatment period.

ELIGIBILITY:
Inclusion Criteria:

* moderate or severe unipolar depression diagnosed according to criteria of Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5)
* duration of the current episode must be ≥ 6 weeks and ≤ 2 years
* HDRS17 ≥ 18
* mild to moderate treatment resistance according to the Antidepressant Treatment History Form [ATHF-SF]. Treatment resistance is defined as having failed at least one but no more than three adequate antidepressant treatments in this episode
* stable antidepressive medication 4 weeks before treatment or no antidepressive treatment
* no further relevant psychiatric axis-I and/or axis-II disorder except for anxiety disorders (according to DSM-5 and SCID-5-PD)
* no comorbid psychotic symptoms
* ability to give consent

Exclusion Criteria:

* acute suicidality (MADRS item 10 score > 4)
* antiepileptic drugs and/or benzodiazepines corresponding to > 1mg lorazepam / day
* history of brain surgery, significant and clinically relevant brain malformation or neoplasm, head injury, stroke, dementia or other neurodegenerative disorder
* history of seizures
* previous rTMS treatment
* lifetime history of non-response to adequate electroconvulsive therapy (minimum of eight treatments)
* deep brain stimulation
* cardiac pacemakers, intracranial implant, or metal in the cranium
* substance dependence or abuse in the past 3 months (with the exception of tobacco)
* severe somatic comorbidity as judged by the study physician
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Response rate of Montgomery-Asberg Depression Rating Scale (MADRS) | 6 weeks
  MADRS reduction of at least 50% of baseline value after end of treatment period between active combined iTBS / cTBS and the sham condition.
  (rater questionnaire; MADRS raw score ranges between 0 and 60; the higher the score, the more severe depression)

SECONDARY OUTCOMES:
Remission rate after treatment | 6 weeks
  Montgomery-Asberg Depression Rating Scale (MADRS) </= 10 after treatment (rater questionnaire; MADRS raw score ranges between 0 and 60; the higher the score, the more severe depression)
Reduction of raw score: Montgomery-Asberg Depression Rating Scale (MADRS) | 6 weeks
  The reduction of the raw score after treatment will be compared between active TBS and sham TBS (rater questionnaire; range between 0 and 60; higher score indicates higher level of severity)
Reduction of raw score: Hamilton Depression Rating Scale 17 items (HDRS17) | 6 weeks
  The reduction of the raw score after treatment will be compared between active TBS and sham TBS (rater questionnaire; score ranges from 0-53;higher score indicates higher level of severity)
Reduction of raw score: Clinical Global Impression (CGI) | 6 weeks
  The reduction of the raw score after treatment will be compared between active TBS and sham TBS (rater questionnaire; score ranges from 0-7; higher score indicates higher level of severity)
Reduction of raw score: Beck Depression Inventory (BDI-II) | 10 and 18 weeks
  The reduction of the raw score during follow-up will be compared between active TBS and sham TBS (self-rating questionnaire; score ranges from 0-63; higher score indicates higher level of severity)
Reduction of raw score: WHO-5 well-being index | 10 and 18 weeks
  The reduction of the raw score during follow-up will be compared between active TBS and sham TBS (self-rating questionnaire; score ranges from 0-25; lower score indicates higher level of severity)
Work Productivity and Activity Impairment Questionnaire (WPAI) | 6 and 18 weeks
  Functionality will be assessed by Work Productivity and Activity Impairment Questionnaire (WPAI; self-rating questionnaire) at baseline, after treatment period as well as during follow-up; contains 6 questions about the effect of health problems on the ability to work and perform regular activities. Health problems are defined as any physical or emotional problem or symptom. Patients are asked to fill in the blanks or circle a number; there is no overall score;
Frequency of adverse events | 6 weeks
  Comparison of both arms in respect to number of adverse events during treatment period
Deterioration rate after treatment period | 6 weeks
  Deterioration is defined as an increase of MADRS (Montgomery-Asberg Depression Rating Scale) score of 25% compared to baseline score (rater questionnaire; range between 0 and 60; higher score indicates higher level of severity)
Examination of the influence of Childhood Trauma Questionnaire (CTQ) at baseline as possible predictor for change of MADRS | 6 weeks
  It will be examined whether the CTQ can be used for predicting treatment effect, measured by Montgomery-Asberg Depression Rating Scale (MADRS, see above)
Examination of the influence of cognitive performance at baseline as possible predictor for change of MADRS | 6 weeks
  It will be examined whether cognitive performance measured by THINC-Integrated Tool (Thinc-it -tool; includes 4 different test covering different aspects of cognition) at baseline can be used for predicting treatment effect, measured by Montgomery-Asberg Depression Rating Scale (MADRS, see above)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Plewnia, Prof., MD, Principal Investigator — Department of Psychiatry and Psychotherapy, University of Tuebingen
Locations (7):
- Germany (7):
  - Department of Psychiatry, Psychotherapy and Psychosomatics, Medical Faculty, University of Augsburg, Bezirkskrankenhaus Augsburg, Augsburg
  - University of Leipzig, Dept. Psychiatry and Psychotherapy, Leipzig
  - University of Munich, Munich
  - University of Regensburg, Dept. Psychiatry and Psychotherapy, Regensburg
  - University of Tuebingen, Dept Psychiatry and Psychotherapy, Tübingen
  - University of Um, Dept. Psychiatry and Psychotherapy, Ulm
  - University of Wuerzburg, Dept. Psychiatry and Psychotherapy, Würzburg

REFERENCES:
- [Derived] Plewnia C, Brendel B, Schwippel T, Nieratschker V, Ethofer T, Kammer T, Padberg F, Martus P, Fallgatter AJ. Treatment of major depressive disorder with bilateral theta burst stimulation: study protocol for a randomized, double-blind, placebo-controlled multicenter trial (TBS-D). Eur Arch Psychiatry Clin Neurosci. 2021 Oct;271(7):1231-1243. doi: 10.1007/s00406-021-01280-w. Epub 2021 Jun 19. PMID 34146143
- See also: This link is related to the published study protocol — https://link.springer.com/article/10.1007/s00406-021-01280-w